CLINICAL TRIAL: NCT05626465
Title: Identification of Novel Biomarker-s of Abusive Head Trauma on Serum by Proteomics
Brief Title: Biomarker-s of Abusive Head Trauma by Proteomics
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Kim Wiskott, Dre Kim Wiskott, University Hospital, Geneva
Other Study IDs: 2021-01971
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Abuse, Child; Protein Disorder, Blood
Keywords: abusive head trauma; proteomic; biomarker
MeSH Terms: conditions — Blood Protein Disorders | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Abusive Head Trauma (AHT)
  Interventions: Other: Blood test
- Accidental traumatic brain injury
  Interventions: Other: Blood test
- Cranioplasty
  Interventions: Other: Blood test
- Infant malaise without AHT
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Proteomic analyses on serum

SUMMARY:
The aim of our study is to highlight biomarker-s of Abusive Head Trauma by proteomics analyses on the serum of child victims of abuse.

ELIGIBILITY:
Inclusion Criteria:

* Age : 0-2 y.o
* Medical consultation for malaise, seizure (without fever), loss of consciousness, traumatic bain injury, or cranioplasty
* Blood test during medical care
* Accepted informed consent

Exclusion Criteria:

* Refused informed consent
* For control groups : medical history of child abuse
* For AHT group : rare metabolic disease (Menkes, etc..)

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infant between 0 to 2 y.o
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Highlight novel biomarker-s of AHT | Hospital admission to discharge (up to 3 days)
  Proteomic analyses will be made on serum of infant victim of AHT. Results will be compare with control groups (traumatic brain injury, cranioplasty, malaise).

CONTACTS AND LOCATIONS:
Overall Officials: Tony Fracasso, Prof., Study Director — University Hospital, Geneva
Locations (2):
- Ginhoux Thiphanie, Lyon, Rhône, France
- Wiskott Kim, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No